CLINICAL TRIAL: NCT05849090
Title: Pilot for Vancomycin and Tobramycin Powder Use in Acute Open Fractures in the Emergency Department
Brief Title: Vancomycin and Tobramycin Powder Use in Acute Open Fractures
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Justin Haller, Principle Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 158712
Record Dates: First submitted 2023-04-11; First posted 2023-05-08 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Infections
Keywords: Infections; Acute open fractures; Standard of care prophylactic antibiotics; Vancomycin and Tobramycin powder
MeSH Terms: conditions — Infections | interventions — Cephalosporins; Clindamycin; Cefazolin; Ceftriaxone; clindamycin phosphate; Vancomycin; Tobramycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care prophylactic antibiotics (Active Comparator): Standard irrigation and IV, cephalosporin, 2-grams, intravenous (IV),
  * or standard irrigation and IV, clindamycin (900mg) / vancomycin (20mg/kg), intravenous (IV) for patients with cephalosporin allergies.
  Interventions: Drug: Cephalosporin or clindamycin/vancomycin antibiotics..
- Vancomycin and Tobramycin (Experimental): One-time dosage of topical vancomycin (1 gram) and tobramycin (1.2 grams) powder.
  Interventions: Drug: Vancomycin and Tobramycin antibiotics.

INTERVENTIONS:
Drug: Cephalosporin or clindamycin/vancomycin antibiotics.. — Antibiotics: Cephalosporin, 2-grams, intravenous (IV), or clindamycin (900mg) / vancomycin (20mg/kg), intravenous (IV).
  Other Names: Cephalosporin - Cefazolin, (Ancef, Kefzol, Cefacidil); Cephalosporin- Ceftriaxone, (Ceftrisol Plus, Rocephin); Clindamycin, (Cleocin, Clindesse); Vancomycin, (Vancocin)
  Arms: Standard of care prophylactic antibiotics
Drug: Vancomycin and Tobramycin antibiotics. — Vancomycin (1 gram) and tobramycin (1.2 grams).
  Other Names: Vancomycin, (Vancocin); Tobramycin, (Tobi, Tobrex, Nebcin)
  Arms: Vancomycin and Tobramycin

SUMMARY:
The investigators overall aim of this study is to determine the difference in 6-month infection rates in patients treated with the combined vancomycin and tobramycin (VT) powder compared to the standard of care (SC).

In order to evaluate this objective, the investigators propose the following specific aims for the pilot study:

Specific Aim 1: Assess VT and SC patient enrollment, randomization and early clinical follow-up. Hypothesis: This study will successfully enroll and randomize 50 patients, 25 into each treatment group and will achieve 85% clinical follow-up at 6-months post-ED admission date.

Open fracture patients/families that meet study inclusion/exclusion criteria will be approached by a study team member for informed consent. After providing consent, patients will be appropriately randomized to either VT or SC treatment. Patients will be clinically followed at regular intervals up to 6 months post-surgery. Enrollment, appropriate randomization and surgical allocation, and clinical follow-up will be evaluated.

Specific Aim 2: Compare infection rates, cultures and patient characteristics between groups. Hypothesis: VT will have a lower infection rate than the SC group. Additionally, randomization will create an equal distribution of patient demographics as well as fracture severity and soft tissue damage, as classified by the Gustilo-Anderson Classification System (GA).

Specific Aim 3: Compare local wound healing and fracture healing between VT group and SC group. Hypothesis: VT will have less rates of wound healing complications due to decreased infections. No local wound irritation or wound closure issues will be seen between groups. There will be no difference in fracture healing between groups.

DETAILED DESCRIPTION:
Open limb fractures are severe orthopedic injuries and at an increased risk for complications including nonunion and infection. Rates of infection are dependent upon features such as extent of soft tissue trauma, patient characteristics, degree of contamination and modifiable factors such as time to surgical debridement and IV (intravenous) antibiotics. Surgical debridement within 24 hours and IV antibiotics are the current standard of care, but despite advances in care, the infection rates for these injuries has remained stable over the last several decades.

Possible explanations for this stagnation in care may be related to the current standard of care and the pathophysiology of open fractures. There is significant soft-tissue damage in open fractures, which compromises local vasculature leading to devascularized soft tissue and bone. This devitalized tissue serves as a nidus for infection, a base for biofilm production and reduces the level of systemic antibiotics delivered to the zone of injury. Local antibiotic therapy has the potential to overcome these challenges, by allowing a high concentration of antibiotics to be delivered to the devitalized tissue. Additional benefits of local antibiotics are their powdered form, which is stable, easy to transport, and can be applied immediately in austere situations without the need for IV access. A recent randomized control trial found a 4% decrease risk of infection following powdered vancomycin placement at the time of hardware fixation. However, a recent meta-analysis showed nearly a 12% risk reduction in open fractures treated with local antibiotics when compared to the standard of care. However, this meta-analysis was predominantly made up of small retrospective studies, underlying the need for a randomized control trial evaluating the efficacy of local antibiotics in acute open fracture management.

While causative organisms vary with location, cultures from open fractures are positive 83% of the time. Cultures have shown high rates of colonization of both gram-positive organisms (predominantly Staphylococcus aureus and epidermidis) as well as gram-negative organisms (mostly Pseudomonaonas aeruginosa). Given this prevalence the antibiotics vancomycin and tobramycin are likely good candidates given that they have high efficacy against the common colonizing bacteria, are available in standardize powdered formula, reach high local concentrations, and have a minimal cytotoxic effect to local cells6. Using a combination of vancomycin and tobramycin in the acute care of severe open fractures may substantially decrease risks of infection from both gram-positive and gram-negative pathogens.

ELIGIBILITY:
Inclusion Criteria:

* Open fracture GA class II or III, and one of the following fracture locations:
* Calcaneus fracture,
* Tibial plafond (pilon) fracture,
* Tibial plateau fracture,
* Tibial shaft fracture,
* Distal femur fracture,
* Femoral shaft fracture.
* Informed consent can be obtained from the patient.
* Consent will be obtained in the Emergency Department.

Exclusion Criteria:

* Known allergy to vancomycin or tobramycin.
* Known kidney disease prior to admission, chronic Kidney Disease stage 4 -5.
* Any patients, family members, or staff who refuse to participate.
* Pregnant women, as identified through pregnancy test which is taken in the emergency department as standard of care.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Percent (%) positive deep tissue infections. | 6-months post-operative
  Percent (%) of positive deep tissue infections (number of infections/total participants X 100).
Percent (%) negative deep tissue infections. | 6-months post-operative
  Percent (%) of negative deep tissue infections (number of infections/total participants X 100).

CONTACTS AND LOCATIONS:
Overall Officials: Justin Haller, M.D., Principal Investigator — University of Utah Orthopaedics
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No